CLINICAL TRIAL: NCT02015767
Title: Patient Registry of Roflumilast In Real Life
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: RO-2455-407-RD; U1111-1146-5619 (Other: WHO Unique Trial Number)
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Drug therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Roflumilast: Participants prescribed roflumilast (Daxas®) according to local guidelines and marketing authorization.

SUMMARY:
A patient registry to capture real life data and demonstrate the performance of roflumilast (Daxas®) in a standard clinical practice.

DETAILED DESCRIPTION:
The drug being tested in this observational study design is called roflumilast, but not as an therapeutic intervention. Roflumilast is approved for and marketed globally for maintenance treatment of severe Chronic Obstructive Pulmonary Disease (COPD) associated with chronic bronchitis in adult patients with a history of frequent exacerbations as add on to bronchodilator treatment.

This study will capture real life data and demonstrate the performance of roflumilast in a standard clinical practice. The study will enroll approximately 1350 (EU)+600(North Asia) patients. This multi-centre trial will be conducted in at least 4 EU and 2 North Asian countries.

The overall time to participate in this study is 12 months. No visits, diagnostic procedures or monitoring will take place, which would not happen had the patient not been included in the study.

Participants will be followed according to usual practice and data recorded approximately at 6 months and at 12 months of roflumilast treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to the data collection
* Roflumilast (Daxas®) treatment initiated in Roflumilast (Daxas®) naïve patients at the time of registry

Exclusion Criteria:

There are no exclusion criteria per se. However it is expected that patients are treated according to locally approved marketing authorisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants prescribed roflumilast (Daxas®) according to local guidelines and marketing authorization.
  The registry sites will comprise hospitals, and office-based physicians. The investigators will be mainly pulmonologists, or as per the standard practice of the specific country.
Sampling Method: Non-Probability Sample
Enrollment: 1950 (Estimated)
Dates: Start 2013-02-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Number of observed exacerbations | 12 months
  Number of exacerbations observed during the study period and per patient per year

SECONDARY OUTCOMES:
Severity of exacerbations | 12 months
  Severity of exacerbations (proportion of exacerbations requiring systemic corticosteroid treatment and/or antibiotics or requiring hospitalization).
Seasonal variation of exacerbation | 12 months
  Seasonal variation of exacerbation during Roflumilast treatment.
Number of hospitalizations due to COPD exacerbations | 12 months
  Number of hospitalizations due to Chronic obstructive pulmonary disease (COPD) exacerbations per patient per year.
Change from Baseline in lung function parameters (FEV1 and FEV1/FVC) | Baseline and Month 12
  Change in lung function parameters parameters FEV1(Forced Expired Volume measured after 1 second expiration) and FEV1/FVC (Forced Vital Capacity) from Baseline to the last recorded value and to the end of the study.
Change from Baseline in blood oxygen saturation | Baseline and Month 12
  Change in blood oxygen saturation assessed with pulse oximetry from Baseline to the last recorded value and the end of the study.
Percentage of compliance to treatment | 12 months
  Estimated percentage of prescribed doses taken since the last date of data collection.
Changes in concomitant administration of COPD maintenance treatments | 12 months
  Changes in concomitant administration of COPD maintenance treatments since start of roflumilast treatment.
Health status using the COPD Assessment Questionnaire (CAT) | Baseline, Month 6 and Month 12
Change from Baseline in breathlessness | Baseline and Month 12
  Change in breathlessness assessed using the Modified Medical Research Council (mMRC) dyspnoea scale, from Baseline to the end of observation.
Number of Participants with adverse Drug Reactions (ADRs) | 12 months
  An ADR is a response to an observed medicinal product which is noxious and unintended resulting not only from the authorised use of a medicinal product at normal doses, but also from medication errors and uses outside the terms of the marketing authorisation, including the misuse and abuse of the medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (51):
- Bulgaria (5):
  - Pleven
  - Razgrad
  - Sofia
  - Troyan Municipality
  - Vratsa
- Greece (16):
  - Agrinio
  - Athens
  - Edessa
  - Herakleion-Crete
  - Imitos
  - Kaisarianí
  - Kalamaria
  - Katerini
  - Nafpaktos
  - Pátrai
  - Peristeri
  - Piraeus
  - Ptolemaida
  - Pýrgos
  - Thessaloniki
  - Volos
- Hong Kong, Hong Kong
- Norway (9):
  - Arendal
  - Bergen
  - Elverum
  - Fredrikstad
  - Kongsvinger
  - Sandvika
  - Skien
  - Straume
  - Tønsberg
- Slovakia (14):
  - Banská Bystrica
  - Bardejov
  - Bratislava
  - Humenné
  - Malacky
  - Michalovce
  - Nitra
  - Považská Bystrica
  - Prešov
  - Revúca
  - Senica
  - Spišská Nová Ves
  - Štúrovo
  - Topoľčany
- South Korea (6):
  - Busan
  - Daegu
  - Gwangju
  - Jeonju
  - Seoul
  - Suwon

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4568&filename=PROFILE%20EU%20Synopsis.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4568&filename=PROFILE%20Asia%20Synopsis.pdf